CLINICAL TRIAL: NCT00666952
Title: Randomized Trial of a Patient Decision Aid for Bariatric Surgery
Brief Title: Study Testing Patient Decision Tools Related to the Risks and Benefits of Weight Loss Surgery
Acronym: POINT of View
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Foundation for Informed Medical Decision Making (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FIMDM IIG Grant 0094-1
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Obesity, Morbid; Obesity; Decision Aids; Bariatric Surgery
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Other: Video Decision Aid
- 2 (Active Comparator)
  Interventions: Other: Booklet Decision Aid

INTERVENTIONS:
Other: Video Decision Aid — Participants randomized to the video decision aid group will be asked to view the video portion of the decision aid, Weight loss surgery: Is it right for you? in a private room The content of the video and accompanying booklet was based on a systematic-review of the efficacy and safety of bariatric surgery, input from experts in bariatric surgery, internal medicine, psychology, nutrition, and nursing, and from a series of focus groups and interviews with 30 morbidly obese patients, some of whom had elected not to have bariatric surgery.
  Arms: 1
Other: Booklet Decision Aid — General educational booklet on gastrointestinal surgery developed by the NIH titled, 'Gastrointestinal Surgery for Severe Obesity'.
  Arms: 2

SUMMARY:
Morbid obesity currently affects more than 11 million US adults and is strongly associated with type 2 diabetes, cancer, cardiovascular disease, and arthritis. Bariatric (weight loss) surgical procedures have been shown to significantly reduce body weight and improve the health and quality of life of morbidly obese adults, at least in the short term. However, bariatric surgery also presents substantial risks, including a 10% to 20% risk of serious complications and up to a 2% risk of death in the first 30 days after surgery. Thus, a morbidly obese patient's decision regarding bariatric surgery should be based on his or her evaluation of accurate information on the possible risks and benefits of the various treatment options. Anecdotal reports suggest that bariatric treatment decisions may be more heavily influenced by insurance coverage and reimbursement rates than patient preferences.

The main objective of the current proposal is to examine the impact of a bariatric decision aid, Weight loss surgery: Is it right for you?, on decision quality in primary care and bariatric specialty practice settings. We propose a randomized controlled trial to assess the effect of this bariatric decision aid on bariatric-specific measures of patient knowledge, values and choice of weight management strategy. We will also investigate the effect of the decision aid on decisional conflict and decisional self-efficacy and examine medical, psychological, and behavioral factors as mediators and moderators of treatment choice. This information will help to elucidate the value of this decision aid in improving decision quality.

The primary aims of this of this research are to:

1. Determine if the bariatric decision aid results in superior bariatric surgery decision quality than an NIH booklet on weight loss surgery ('usual care').
2. Determine if the bariatric decision aid results in less decisional conflict and superior decisional self-efficacy than usual care.
3. Determine if there is a differential effect of the interventions on decision quality among treatment seekers and non-treatment seekers.
4. Investigate medical, psychological, and behavioral factors as mediators of treatment choice.

The secondary aims of this study are to:

1. Understand the current weight control attitudes and practices among morbidly obese patients who are not actively seeking bariatric surgical treatment.
2. Assess the rates of bariatric surgery, health care costs, health care use and outcomes, and changes in BMI over time across the intervention groups, as well as across study subgroups, such as those who did and did not choose to have bariatric surgery.

We hypothesize that the decision aid will result in greater knowledge and greater values concordance, less decisional conflict and superior decisional self-efficacy than the NIH booklet.

ELIGIBILITY:
Inclusion Criteria:

* aged 20 to 65 years
* enrolled in Group Health and not planning to discontinue enrollment during study period
* meet standard NIH eligibility criteria for bariatric surgery
* reside in King County;
* have a phone
* are able to read, write and speak in English
* report no physical or hearing impairments which would prevent engaging in the study assessments

Exclusion Criteria:

* Pregnant, lactating, or planning to become pregnant in the next two years
* have any contraindications to bariatric surgery
* previously undergone a bariatric procedure

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Our primary focus is estimating the benefit of the decision aid on decision quality. The two components of decision quality are knowledge and value concordance. | 3 Months

SECONDARY OUTCOMES:
Our secondary aims will examine the impact of our interventions or decisional conflict, decisional self-efficacy, and explore potential mediators of our intervention effects. | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: David E Arterburn, MD, MPH, Principal Investigator — Group Health Research Institute
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States